CLINICAL TRIAL: NCT03689010
Title: A Multi-Center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group Study, Comparing Taro Product to RLD, and Both Active Treatments to a Placebo Control in the Treatment of Moderate Facial Rosacea
Brief Title: To Evaluate the Therapeutic Equivalence and Safety in Treatment of Moderate Facial Rosacea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AZAF-1703
Record Dates: First submitted 2018-09-21; First posted 2018-09-28 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — azelaic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Azelaic acid foam 15% (Active Comparator): Topical, twice daily (Apply the foam (morning and evening) to the entire facial area (cheeks, chin, forehead, and nose).
  Interventions: Drug: Azelaic acid foam 15%
- Finacea® (azelaic acid) Foam, 15% (Active Comparator): Topical, twice daily (Apply the foam (morning and evening) to the entire facial area (cheeks, chin, forehead, and nose).
  Interventions: Drug: Finacea® (Azelaic acid Foam) 15%
- Vehicle of the test product (Placebo Comparator): Topical, twice daily (Apply the foam (morning and evening) to the entire facial area (cheeks, chin, forehead, and nose).
  Interventions: Drug: Vehicle of the test product

INTERVENTIONS:
Drug: Azelaic acid foam 15% — Azelaic acid foam 15%
  Other Names: AZAF 1703
  Arms: Azelaic acid foam 15%
Drug: Finacea® (Azelaic acid Foam) 15% — Azelaic acid foam 15%
  Arms: Finacea® (azelaic acid) Foam, 15%
Drug: Vehicle of the test product — Vehicle of the test product
  Other Names: Placebo
  Arms: Vehicle of the test product

SUMMARY:
To demonstrate the superiority of the efficacy of the test and reference products over that of the placebo control in the treatment of moderate facial rosacea.

DETAILED DESCRIPTION:
A Multi-Center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group study, comparing test and reference products and both active treatments to a placebo control in the treatment of Moderate Facial Rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female aged ≥ 18 with a clinical diagnosis of facial rosacea.
* Subjects must have provided IRB approved written informed consent.

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.
* Subjects who have used estrogens or oral contraceptives for less than 3 months prior to baseline; use of such therapy must remain constant throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
change in the inflammatory lesion counts | 12 weeks
  Percent change from baseline to Week 12 in the inflammatory (papules and pustules) lesion counts

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Yantovskiy, Study Director — Taro Pharmaceuticals
Locations (1):
- Catawba Research, LLC, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No